CLINICAL TRIAL: NCT02093897
Title: A Phase III Open-label Pharmacokinetic, Efficacy and Safety Study of rVIII-SingleChain in a Pediatric Population With Severe Hemophilia A
Brief Title: Pharmacokinetic, Efficacy, and Safety Study of Recombinant Factor VIII Single Chain (rVIII-SingleChain) in Children With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL627_3002; 2012-001336-65 (EudraCT Number)
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Congenital Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rVIII-SingleChain (Experimental): Subjects will be assigned to either an on-demand or prophylaxis regimen and will receive rVIII-SingleChain as an intravenous (IV) infusion. Subjects assigned to a prophylaxis regimen will be treated with 15 to 50 IU/kg of rVIII-SingleChain every second day or 2 to 3 times per week, or at the investigator's discretion, based on available PK data, the FVIII treatment regimen used before enrollment and/or the subject's bleeding phenotype. The dose for on-demand treatment of a bleeding episode is based on the recommendations of the World Federation of Hemophilia (WFH), with a minimum dose of 15 IU/kg. All subjects were to be treated for a minimum of 50 EDs. For the PK evaluation, the subjects will receive a single IV dose of 50 IU/kg of rVIII-SingleChain on Day 1 at the start of the PK evaluation period.
  Interventions: Biological: rVIII-SingleChain

INTERVENTIONS:
Biological: rVIII-SingleChain
  Other Names: Recombinant Factor VIII single chain; CSL627

SUMMARY:
This is an international, multicenter, open-label study to assess the efficacy, safety, and pharmacokinetic (PK) profile of rVIII-SingleChain in pediatric patients with severe hemophilia A. A minimum of 25 previously treated subjects ≥ 6 to < 12 years of age and at least 25 subjects < 6 years of age who have undergone > 50 exposure days (EDs) with a previous Factor VIII (FVIII) product are planned to be enrolled. Subjects will be assigned to either an on-demand or prophylaxis treatment regimen and will receive rVIII-SingleChain at a dose to be determined by the investigator. Hemostatic efficacy will be assessed by the subject/caregiver and the investigator who will assess overall efficacy by a 4-point scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe hemophilia A defined as < 1% Factor VIII (FVIII) concentration (FVIII:C) documented in medical records,
* Males < 12 years of age,
* Subjects who have received > 50 EDs with a FVIII product,
* Prior PK data (at least incremental recovery and half-life) from previous FVIII exposure for subjects participating in the PK part
* Investigator believes that the subject is willing and able to adhere to all protocol requirements. Investigator believes that the subject's parent(s) or legally acceptable representative(s) is / are willing and able to adhere to all protocol requirements.

Exclusion Criteria:

* Any history of or current FVIII inhibitors
* Use of an Investigational Medical Product (IMP) within 30 days prior to the first rVIII-SingleChain administration,
* Administration of any cryoprecipitate, whole blood or plasma within 30 days prior to administration of rVIII-SingleChain,
* Known hypersensitivity (allergic reaction or anaphylaxis) to any FVIII product or hamster protein,
* Subject currently receiving IV immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment,
* Subject with serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) values >5 times (x) the upper limit of normal (ULN) at Screening,
* Subjects with serum creatinine values >2 x ULN at Screening,
* Evidence of thrombosis, including deep vein thrombosis, stroke, pulmonary embolism, myocardial infarction and arterial embolus within 3 months before Day 1,
* Experienced life-threatening bleeding episode or had major surgery or an orthopedic surgical procedure during the 3 months before rVIII-SingleChain administration.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (36):
- United States (2):
  - Study Site, Aurora, Colorado
  - Study Site, Chicago, Illinois
- Study Site, Melbourne, Victoria, Australia
- Austria (2):
  - Study Site, Linz
  - Study Site, Vienna
- France (5):
  - Study Site, Brest
  - Study Site, Le Kremlin-Bicêtre
  - Study Site, Lille
  - Study Site, Nantes
  - Study Site, Paris
- Study Site, Tbilisi, Georgia
- Germany (4):
  - Study Site, Bonn
  - Study Site, Bremen
  - Study Site, Frankfurt am Main
  - Study Site, Hanover
- Study Site, Milan, Italy
- Study Site, Beirut, Lebanon
- Study Site, Kuala Lumpur, Malaysia
- Netherlands (3):
  - Study Site, Amsterdam
  - Study Site, Njmegen
  - Study Site, Utrecht
- Philippines (2):
  - Study Site, Cebu City
  - Study Site, Davao City
- Study Site, Rzeszów, Poland
- Study Site, Porto, Portugal
- Study Site, Timișoara, Romania
- Study Site, Madrid, Spain
- Study Site, Lucerne, Switzerland
- Thailand (4):
  - Study Site, Bangkok
  - Study Site, Chiang Mai
  - Study Site, Khon Kaen
  - Study Site, Songkhla
- Turkey (Türkiye) (3):
  - Study Site, Adana
  - Study Site, Istanbul
  - Study Site, Izmir
- Study Site, Lviv, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, multinational study enrolled subjects at 37 participating study centers in Australia, Europe, Georgia, Lebanon, Malaysia, Philippines, Switzerland, Thailand, Turkey, Ukraine, and the United States.
Pre-assignment Details: Screening took place 4 to 28 days prior to first dose of study product (rVIII-SingleChain). A total of 88 subjects were screened, 4 of these did not fulfill all eligibility criteria and were therefore screening failures.
Groups:
- rVIII-SingleChain: Subjects were assigned to either an on-demand or prophylaxis regimen and received rVIII-SingleChain as an intravenous (IV) infusion. Subjects assigned to a prophylaxis regimen were treated with 15 to 50 IU/kg of rVIII-SingleChain every second day or 2 to 3 times per week, or at the investigator's discretion, based on available PK data, the FVIII treatment regimen used before enrollment and/or the subject's bleeding phenotype. The dose for on-demand treatment of a bleeding episode was based on the recommendations of the World Federation of Hemophilia (WFH), with a minimum dose of 15 IU/kg. All subjects were to be treated for a minimum of 50 EDs. For the PK evaluation, the subjects received a single IV dose of 50 IU/kg of rVIII-SingleChain on Day 1 at the start of the PK evaluation period.
Period: Overall Study
Arm/Group | rVIII-SingleChain
Started (A total of 5313 CSL627 infusions were administered to 84 subjects during the study.) | 84
Completed (As planned, groups were closed and subjects discontinued when 25 subjects reached 50 EDs per group.) | 65
Not Completed | 19
Not completed — Physician Decision | 1
Not completed — Planned age group closure - no's reached | 17
Not completed — Adverse event, non-fatal | 1

BASELINE CHARACTERISTICS:
Groups:
- rVIII-SingleChain: Subjects were assigned to either an on-demand or prophylaxis regimen and received rVIII-SingleChain as an IV infusion. Subjects assigned to a prophylaxis regimen were treated with 15 to 50 IU/kg of rVIII-SingleChain every second day or 2 to 3 times per week, or at the investigator's discretion, based on available PK data, the FVIII treatment regimen used before enrollment and/or the subject's bleeding phenotype. The dose for on-demand treatment of a bleeding episode was based on the recommendations of the WFH, with a minimum dose of 15 IU/kg. All subjects were to be treated for a minimum of 50 EDs. For the PK evaluation, the subjects received a single IV dose of 50 IU/kg of rVIII-SingleChain on Day 1 at the start of the PK evaluation period.
Arm/Group | rVIII-SingleChain
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (3.11)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 84
Type of FVIII product used before enrollment [Number; unit: participants] — Type of FVIII product used by the subjects within the 12 months before enrollment into the study. This could have been a plasma FVIII product or a recombinant FVIII product.
  participants
    Plasma product | 33
    Recombinant Product | 49
    Unknown | 2
Treatment modality of FVIII therapy before enrollment [Number; unit: participants] — Treatment modality of FVIII therapy within the 12 months before enrollment, ie, routine prophylaxis or on-demand treatment. If a subject used both modalities, only the most recent one was counted.
  participants
    Prophylaxis | 60
    On-Demand | 24

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: Rate of treatment success where treatment success of a bleeding episode is defined as a rating of "excellent" or "good" based on the investigator's overall clinical assessment of hemostatic efficacy (using a 4-point scale of excellent, good, moderate or poor/no response) on the on-demand and prophylaxis regimens combined. The rate of success was based on the number of treated bleeding events; there were 347 treated bleeding events in the Efficacy Population.
Time Frame: Up to 1 year
Population: Efficacy Population
Measure: Number (95% Confidence Interval); unit: Percentage of treated bleeding events
Units Other Than Participants: Treated bleeding events
Groups:
- Efficacy Population: The Efficacy Population consisted of all subjects who received at least 1 dose of rVIII-SingleChain as part of either a routine prophylaxis or on-demand regimen during the study. One subject was excluded from the efficacy population because of a pre-existing inhibitor to FVIII (confirmed by reexamination of a screening sample initially reported as negative due to laboratory error).
Arm/Group | Efficacy Population
Number analyzed (Participants) | 83
Number analyzed (Treated bleeding events) | 347
Percentage of treated bleeding events | 96.3 [91.3 to 98.4]

2. Secondary Outcome: Annualized Bleeding Rate
Description: The annualized bleeding rate was defined as the number of bleeding episodes requiring treatment divided by the efficacy evaluation period in days, x 365.25, and is presented separately for the on-demand regimen and the prophylaxis regimens.
Time Frame: Up to 1 year
Population: The Efficacy Population comprised all subjects who received at least 1 rVIII-SingleChain dose for prophylaxis or on-demand treatment. One subject was excluded from the efficacy population because of a pre-existing inhibitor to FVIII (confirmed by reexamination of a screening sample initially reported as negative due to laboratory error).
Measure: Median (Inter-Quartile Range); unit: Treated bleeding episodes per year
Groups:
- On-demand: Subjects assigned to the on-demand treatment regimen treated themselves, or were treated by a caregiver/guardian, as needed for any bleeding episode and did not receive routine assigned infusions.
- Prophylaxis: Subjects receiving routine prophylaxis treatment were initially treated with 15-50 IU/kg of rVIII-SingleChain every second day or 2 to 3 times per week, or at the investigator's discretion, based upon available PK data, the FVIII treatment regimen used before enrollment and/or the subject's bleeding phenotype. The dose or dosing frequency may have been adjusted if necessary.
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 3 | 80
Treated bleeding episodes per year | 78.56 [35.12 to 86.62] | 3.69 [0.00 to 7.20]

3. Secondary Outcome: Percentage of Bleeding Episodes Requiring 1, 2, 3, or More Than 3 Infusions of rVIII-SingleChain to Achieve Hemostasis.
Time Frame: Up to 1 year
Population: Efficacy Population
Measure: Number; unit: Percentage (%) of bleeding episodes
Units Other Than Participants: Number of Treated Bleeds
Arm/Group | Efficacy Population
Number analyzed (Participants) | 83
Number analyzed (Number of Treated Bleeds) | 347
Percentage (%) of bleeding episodes
  Requiring 1 infusion | 85.9
  Requiring 2 infusions | 9.8
  Requiring 3 infusions | 2.3
  Requiring > 3 infusions | 2.0

4. Secondary Outcome: Consumption of rVIII-SingleChain - IU/kg Per Subject Per Month
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Median (Full Range); unit: IU/kg per subject per month
Groups:
- On-demand: Subjects assigned to the on-demand treatment regimen treated themselves, or were treated by a caregiver/guardian, as needed for any bleeding episode and did not receive routine assigned infusions. Preventative and additional doses of rVIII-SingleChain were allowed. "Preventative dose" was defined as a dose taken before an activity or a minor procedure to prevent or minimize a bleeding episode, and "additional dose" was defined as a dose taken beyond the need to control hemostasis.
- Prophylaxis: Subjects receiving routine prophylaxis treatment were initially treated with 15-50 IU/kg of rVIII-SingleChain every second day or 2 to 3 times per week, or at the investigator's discretion, based upon available PK data, the FVIII treatment regimen used before enrollment and/or the subject's bleeding phenotype. The dose or dosing frequency may have been adjusted if necessary. Preventative and additional doses of rVIII-SingleChain were allowed. "Preventative dose" was defined as a dose taken before an activity or a minor procedure to prevent or minimize a bleeding episode, and "additional dose" was defined as a dose taken beyond the need to control hemostasis.
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 3 | 80
IU/kg per subject per month | 202 [126 to 231] | 378 [153 to 1394]

5. Secondary Outcome: Consumption of rVIII-SingleChain - IU/kg Per Subject Per Year
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Median (Full Range); unit: IU/kg per subject per year
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 3 | 80
IU/kg per subject per year | 2429 [1508 to 2771] | 4541 [1839 to 16727]

6. Secondary Outcome: Consumption of rVIII-SingleChain - IU/kg Per Bleeding Event
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Median (Full Range); unit: IU/kg per event
Arm/Group | On-demand | Prophylaxis
Number analyzed (Participants) | 3 | 80
IU/kg per event | 25.9 [21 to 78] | 37.0 [16 to 282]

7. Secondary Outcome: Consumption of rVIII-SingleChain (On-demand Regimen) - Number of Infusions Per Subject Per Month
Time Frame: Up to 1 year
Population: Subjects assigned to the on-demand treatment regimen.
Measure: Median (Full Range); unit: number of infusion per subject per month
Arm/Group | On-demand
Number analyzed (Participants) | 3
number of infusion per subject per month | 7.58 [5.1 to 7.7]

8. Secondary Outcome: Consumption of rVIII-SingleChain (On-demand Regimen) - Number of Infusions Per Subject Per Year
Time Frame: Up to 1 year
Population: Subjects assigned to the on-demand treatment regimen.
Measure: Median (Full Range); unit: number of infusions per subject per year
Arm/Group | On-demand
Number analyzed (Participants) | 3
number of infusions per subject per year | 90.95 [60.9 to 92.3]

9. Secondary Outcome: Incremental Recovery
Description: Incremental recovery expressed as (IU/dL)/(IU/kg) corrected for subject's predose plasma FVIII activity measured using the chromogenic substrate assay.
Time Frame: At 1 hour after the start of infusion
Population: PK Population
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Groups:
- Pharmacokinetic Population: The Pharmacokinetic (PK) Population comprised those subjects who participated in the PK assessment and received at least 1 dose of rVIII-SingleChain and for whom a sufficient number of analyzable PK samples were obtained to permit the evaluation of the PK profile of rVIII-SingleChain.
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 39
(IU/dL)/(IU/kg) | 1.63 (0.329)

10. Secondary Outcome: Half-life (t1/2) of rVIII-SingleChain
Description: Half-life (t1/2) of rVIII-SingleChain, baseline uncorrected; plasma FVIII activity measured using the chromogenic substrate assay.
Time Frame: Immediately before dosing, and at approximately 1, 5, 10, 24, and 48 hours after dosing.
Population: PK Population
Measure: Mean (Standard Deviation); unit: hour
Groups:
- Pharmacokinetic Population: The PK Population comprised those subjects who participated in the PK assessment and received at least 1 dose of rVIII-SingleChain and for whom a sufficient number of analyzable PK samples were obtained to permit the evaluation of the PK profile of rVIII-SingleChain.
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 39
hour | 10.3 (2.51)

11. Secondary Outcome: Area Under the Concentration Curve (AUC)
Description: AUC to the last sample with quantifiable drug concentration (AUC0-t), baseline uncorrected; plasma FVIII activity measured using the chromogenic substrate assay.
Time Frame: Immediately before dosing, and at approximately 1, 5, 10, 24, and 48 hours after dosing.
Population: PK Population
Measure: Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 39
IU*h/dL | 1050 (286)

12. Secondary Outcome: Clearance (Cl) of rVIII-SingleChain
Description: Clearance (Cl) of rVIII-SingleChain, baseline uncorrected; plasma FVIII activity measured using the chromogenic substrate assay.
Time Frame: Immediately before dosing, and at approximately 1, 5, 10, 24, and 48 hours after dosing.
Population: PK Population
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 39
mL/h/kg | 4.86 (1.43)

13. Secondary Outcome: Number of Subjects With Inhibitor Formation to rVIII-SingleChain
Description: The number of subjects who develop inhibitors to rVIII-SingleChain, defined as a rVIII-SingleChain antibody titer of at least 0.6 Bethesda Units (BU) per mL after receiving study drug.
Time Frame: At screening, then after dosing at approximately monthly intervals for 6 months, then every 3 months until reaching 50 EDs, and at the end of study visit (up to approximately 12 months).
Measure: Number; unit: participants
Arm/Group | rVIII-SingleChain
Number analyzed (Participants) | 84
participants | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, approximately 1 year, 5 months.
Description: The Safety Population comprised all subjects treated with rVIII-SingleChain. A total of 5313 CSL627 infusions were administered to 84 subjects during the study.
Arm/Group | rVIII-SingleChain
Serious Adverse Events (participants affected / at risk) | 9/84
Other Adverse Events (participants affected / at risk) | 31/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rVIII-SingleChain (N=84)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Inhibiting antibodies positive (Investigations) | 1 (1) — Subject identified with pre-existing inhibitor to FVIII confirmed by reexamination of screening sample initially reported as negative due to laboratory error. Therefore, event is not a de-novo inhibitor developed during exposure to rVIII-SingleChain
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Device occlusion (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rVIII-SingleChain (N=84)
Head injury (Injury, poisoning and procedural complications) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Headache (Nervous system disorders) | 7 (9)
Pyrexia (General disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Nasopharyngitis (Infections and infestations) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.